CLINICAL TRIAL: NCT04668872
Title: Correlation of Histopathological Findings With Radiation Exposure Levels After Y90 Transarterial Radioembolization (TARE) of Hepatic Metastases: A Feasibility Study
Brief Title: Biopsy After Radioembolization to Identify Changes in Tumor Cells From the Radiation
Status: Recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 20-355
Record Dates: First submitted 2020-12-09; First posted 2020-12-16 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Colon Cancer Liver Metastasis; Colon Cancer; Adenocarcinoma of the Colon; Adenocarcinoma of the Rectum; Liver Metastasis Colon Cancer; Colorectal Cancer
Keywords: colorectal liver metastases; transarterial radioembolization; Y90 TARE; Colon Cancer Liver Metastasis; Colon Cancer; Adenocarcinoma of the Colon; Adenocarcinoma of the Rectum; Colorectal Cancer; Memorial Sloan Kettering Cancer Center; 20-355
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms; Colorectal Neoplasms | interventions — Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with colorectal cancer liver metastases: The study population is represented by patients with colorectal cancer liver metastases that have been deemed clinically appropriate/eligible to receive Y90 TARE for the management of their liver metastases.
  Interventions: Radiation: Y90 TARE; Diagnostic Test: PET/CT; Diagnostic Test: PET/MRI

INTERVENTIONS:
Radiation: Y90 TARE — Y90 TARE will be performed as standard of care (SOC)/clinically indicated: 1) in a lobar or sub-lobar fashion (depending on tumor involvement and location; also targeting the tumor as selective as possible and sparing as much as possible of non-involved liver parenchyma), for participants with extensive bilobar disease or 2) in a radiation segmentectomy approach, intending to deliver 190 Gy radiation dose to target tumor: for patients with limited liver metastatic disease, not amenable for surgery or ablation.
  Other Names: 90Y transarterial radioembolization
Diagnostic Test: PET/CT — Following 90Y TARE, participants will receive a PET/CT or PET/MRI scan to measure the dose administered to the target tumor(s) and uninvolved hepatic parenchyma.
Diagnostic Test: PET/MRI — Following 90Y TARE, participants will receive a PET/CT or PET/MRI scan to measure the dose administered to the target tumor(s) and uninvolved hepatic parenchyma.

SUMMARY:
The purpose of this study is to study the way radioembolization works by collecting biopsy samples of participants' tumors after the procedure. This research may improve the way that radioembolization is performed, which could help people whose cancer has spread to the liver. The research may also provide information about how tumors respond to radioembolization.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* histologically confirmed primary adenocarcinoma of the colon or rectum
* CLM considered unresectable or not amenable to percutaneous ablation
* existent tissue samples from a standard of care biopsy of the target tumor within 42 days prior to treatment OR clinical indication for biopsy at the time of the treatment under the institutional guidelines for progression of disease.
* adequate blood cell counts (WBC > 1.5 x 109/L, platelet count > 50 x 109/L)
* adequate renal function (creatinine < 1.5 mg/dL)
* total bilirubin level ≤ 1.5 mg/dL

Additional inclusion criteria for patients, undergoing 90Y radiation segmentectomy:

A. patients not amenable to surgery or thermal ablation

Exclusion Criteria:

Study exclusion criteria will be similar to general TARE exclusion criteria, which are as follows:

* prior hepatic radiotherapy (The lesion / lobe being treated cannot have had prior treatment with radiotherapy - untreated lesions / lobes in the liver may be evaluated under the protocol)
* severe cirrhosis
* severe portal hypertension
* uncorrectable flow to the gastrointestinal tract and/or >30 Gy (or >50 Gy in multiple sessions) radiation absorbed dose to the lungs

All patients with liver-dominant disease will be considered candidates for TARE even in the face of oligometastatic (up to 5 sites) extrahepatic disease, that is stable or controlled by chemotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients will be identified and recruited from the existing patient population in the Interventional Oncology/Radiology Service of the Department of Radiology at Memorial Sloan-Kettering Cancer Center (MSKCC). The patients will be presented with a study consent form and an explanation of any concerns they may have by the Principal Investigator or research team (i.e. Co-Investigators and consenting professionals).
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-12-07 (Actual); Primary Completion 2026-12-07 (Estimated); Study Completion 2026-12-07 (Estimated)

PRIMARY OUTCOMES:
Correlation of tissue necrosis and radiation-induced cell injury levels with delivered dose at 72 hours | 72 hours after treatment
  Determine the feasibility of correlating tissue necrosis and radiation-induced cell injury levels with delivered dose within the target colorectal cancer liver metastases (CLM) and the uninvolved liver parenchyma.
Correlation of tissue necrosis and radiation-induced cell injury levels with delivered dose at 14-21 days | Between 14-21 days after treatment
  Determine the feasibility of correlating tissue necrosis and radiation-induced cell injury levels with delivered dose within the target colorectal cancer liver metastases (CLM) and the uninvolved liver parenchyma.

CONTACTS AND LOCATIONS:
Overall Officials: Constantinos T Sofocleous, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org